CLINICAL TRIAL: NCT00682643
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Multicenter, Two-Year Study to Evaluate the Ocular Safety of Once-Daily, Fluticasone Furoate Nasal Spray 110mcg in Adults and Adolescents 12 Years of Age and Older With Perennial Allergic Rhinitis
Brief Title: A Clinical Study With Fluticasone Furoate Nasal Spray And Vehicle Placebo For The Treatment Of Perennial (Year-round) Allergic Rhinitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FFR110537
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Results first posted 2012-03-13 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2016-11

CONDITIONS: Rhinitis, Allergic, Perennial
Keywords: Perennial Allergic Rhinitis; fluticasone furoate; ocular safety
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- vehicle placebo nasal spray (Placebo Comparator)
  Interventions: Drug: vehicle placebo nasal spray
- fluticasone furoate nasal spray (Active Comparator)
  Interventions: Drug: fluticasone furoate nasal spray

INTERVENTIONS:
Drug: fluticasone furoate nasal spray — fluticasone furoate nasal spray
  Arms: fluticasone furoate nasal spray
Drug: vehicle placebo nasal spray — placebo
  Arms: vehicle placebo nasal spray

SUMMARY:
The purpose of this study is to assess long-term ocular safety of fluticasone furoate nasal spray in adult and adolescent subjects diagnosed with perennial allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for enrollment in the study must meet all of the following criteria:

- Informed consent

* Subject has provided an appropriately signed and dated informed consent. An appropriately signed and dated assent must be obtained from the parents or guardian if the subject is a child under 18 years of age.

  * Outpatient
* Subject is treatable on an outpatient basis.

  * Age
* 12 years of age and older at Visit 2

  * Male or eligible female Female subjects should not be enrolled if they plan to become pregnant during the time of study participation.

To be eligible for entry into the study, females of childbearing potential must commit to the consistent and correct use of an acceptable method of birth control, as defined by the following:

* Abstinence Females of childbearing potential who are not sexually active must commit to complete abstinence from intercourse for two weeks before exposure to the study drug, throughout the clinical trial, and for a period after the trial to account for elimination of the drug (minimum of six days).
* Oral contraceptive (either combined estrogen/progestin or progestin only)
* Injectable progestogen
* Implants of levonorgestrel
* Percutaneous contraceptive patches
* Intrauterine device (IUD) or intrauterine system (IUS) with a documented failure rate of less than 1% per year,
* Male partner who is sterile (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study and is the sole sexual partner for that female subject, or
* Double barrier method-condom or occlusive cap (diaphragm or cervical /vault caps) plus Spermicide,
* Estrogenic vaginal ring. A urine pregnancy test will be done at the screening visit to confirm females of childbearing potential are not pregnant upon entry into the study. In addition, urine pregnancy tests will be done for all females of childbearing potential at each clinic visit.

  * Diagnosis of PAR to include:

A positive skin test (by prick method) response to appropriate perennial allergen (house dust mites, animal dander, mold, or cockroach) within last 12 months prior to Visit 1 or at Visit 1.

A positive skin test is defined as a wheal ³3mm larger than the diluent control for prick testing.

•Two year medical history and past treatment of PAR (written or verbal confirmation) which includes perennial, i.e., year-round, symptoms. PAR symptoms could include nasal congestion, rhinorrhea, nasal itching and sneezing.

In vitro tests for specific IgE (such as RAST, PRIST) will not be allowed for the diagnosis of PAR.

NOTE: Subjects who meet the above criteria and who also may have seasonal allergic rhinitis (SAR) and/or perennial non-allergic rhinitis (PNAR) are eligible for randomization.

* Environment

  •Subject must be symptomatic to appropriate perennial allergen (animal dander, house dust mites, cockroach, mold) and willing to maintain, as much as possible, the same environment throughout the study.
* Ability to comply with study procedures Subject understands and is willing, able and likely to comply with study procedures and restrictions.
* Literate Subject must be able to read, comprehend, and record information in English

Exclusion Criteria:

Subjects meeting any of the following criteria must not be enrolled in the study:

* Significant concomitant medical conditions, defined as but not limited to:

  * A historical or current evidence of clinically significant uncontrolled disease of any body system (e.g., tuberculosis, psychological disorders, eczema). Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through study participation or which would confound the interpretation of the study results if the disease/condition exacerbated during the study.
  * History or current diagnosis of diabetes mellitus
  * Uncontrolled hypertension (i.e., systolic blood pressure ³ 140mm Hg or diastolic blood pressure ³ 90mm Hg)
  * A severe physical obstruction of the nose (e.g., deviated septum or nasal polyp) or nasal septal perforation that could affect the deposition of double blind intranasal study drug
  * Nasal (e.g., nasal septum) or ocular injury/surgery in the last 6 months (including LASIK eye surgery)
  * Asthma, with the exception of mild intermittent asthma [National Asthma Education and Prevention Program (NAEPP) Guidelines for the Diagnosis and Management of Asthma - Expert Panel Report 3, National Institutes of Health, August 28, 2007.

NOTE: Subjects will be allowed to use short-acting inhaled beta2 agonists ONLY on an as needed basis.

* Rhinitis medicamentosa
* Bacterial or viral infection (e.g., common cold) of the eyes or upper respiratory tract within two weeks of Visit 1 or during the screening period
* Documented evidence of acute or significant chronic sinusitis, as determined by the individual investigator
* Current or history of glaucoma and/or ocular herpes simplex
* Current cataract and/or previous history of cataract surgery
* Physical impairment that would affect subject's ability to participate safely and fully in the study
* Clinical evidence of a Candida infection of the nose
* History of psychiatric disease, intellectual deficiency, poor motivation, substance abuse (including drug and alcohol) or other conditions that will limit the validity of informed consent or that would confound the interpretation of the study results
* History of adrenal insufficiency
* History of Hepatitis B or C

  * Use of corticosteroids, defined as:
* Intranasal corticosteroid within 4 weeks prior to Visit 1 (e.g., VERAMYST, FLONASE™, Nasonex, Rhinocort).
* Inhaled, oral, intramuscular, intravenous, ocular, and/or topical corticosteroids (with the exception of topical hydrocortisone, 1% or less, or equivalent) within 8 weeks prior to Visit 1.

  * Use of other allergy medications within the timeframe indicated relative to Visit 1
* Intranasal or ocular cromolyn within 14 days prior to Visit 1 (e.g., Nasalcrom, Crolom)
* Short-acting prescription and non-prescription antihistamines, including ocular preparations and antihistamines contained in insomnia and "night time" pain formulations, within 3 days prior to Visit 1 (e.g., Benadryl, Chlortrimeton, Dimetane, Tavist)
* Long-acting antihistamines within 10 days prior to Visit 1 (e.g., Allegra, Claritin, Clarinex, Zyrtec).
* Intranasal antihistamines (e.g., Astelin) within 2 weeks prior to Visit 1
* Oral or intranasal decongestants within 3 days prior to Visit 1 (e.g., Sudafed)
* Long-acting beta-agonists within 3 days prior to Visit 1 (e.g., SEREVENT™, Foradil)
* Intranasal, oral, or inhaled anticholinergics within 3 days prior to Visit 1 (e.g., Atrovent)
* Oral antileukotrienes within 3 days of Visit 1 (e.g., Singulair)
* Subcutaneous omalizumab (Xolair) within 5 months of Visit 1
* Use of other medications that may affect allergic rhinitis or its symptoms
* Chronic use of concomitant medications, such as tricyclic antidepressants, that would affect assessment of the effectiveness of the study drug
* Use of other intranasally administered medications (e.g., Miacalcin)

  * Use of immunosuppressive medications 8 weeks prior to screening and during the study
  * Immunotherapy Immunotherapy patients may be enrolled in the study if the immunotherapy was not initiated within 30 days of Visit 1, if the dose has remained fixed over the 30 days prior to Visit 1, and the dose will remain fixed for the duration of the study.
  * Use of any medications that significantly alter the pharmacokinetics of fluticasone furoate (ritonavir and ketoconazole)
  * Use of chronic treatment with agents known to promote the development of cataracts (e.g., potassium-sparing diuretics and allopurinol)
  * Allergy/Intolerance
* Known hypersensitivity to corticosteroids or any excipients

  * Clinical trial/experimental medication experience
* Has recent exposure to an investigational study drug within 30 days of Visit 1
* Participation in a previous or current FFNS (GW685698X) clinical study

  * Positive urine pregnancy test or female who is breastfeeding
* Has a positive or inconclusive pregnancy test at Visit 1 or Visit 2

  * Affiliation with investigational site
* Subject is a participating investigator, sub-investigator, study co-ordinator, or employee of a participating investigator, or is an immediate family member of the aforementioned.

  * Tobacco use
* Subject currently uses smoking products including cigarettes, cigars, and pipe or chewing tobacco, or has used these products in the last 6 months

  * Chickenpox or measles A subject is not eligible if he/she currently has chickenpox or measles, or has been exposed to chickenpox or measles during the last three weeks and is non-immune. If a subject develops chickenpox or measles during the study, he/she will be withdrawn from the study. If a non-immune subject is exposed to chickenpox or measles during the study, his/her continuation in the study will be at the discretion of the investigator, taking into consideration the likelihood of developing active disease.
  * Findings of a clinically significant, abnormal ECG
  * Findings of a clinically significant laboratory abnormality

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2008-06; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (52):
- United States (52):
  - GSK Investigational Site, Oxford, Alabama
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Mission Viejo, California
  - GSK Investigational Site, Rolling Hills Estates, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, Stockton, California
  - GSK Investigational Site, Vista, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Englewood, Colorado
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Conyers, Georgia
  - GSK Investigational Site, Gainesville, Georgia
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Stockbridge, Georgia
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, North Dartmouth, Massachusetts
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Bozeman, Montana
  - GSK Investigational Site, Bellevue, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Ocean City, New Jersey
  - GSK Investigational Site, Skillman, New Jersey
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Sylvania, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Summerville, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, Kerrville, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Waco, Texas
  - GSK Investigational Site, South Burlington, Vermont
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Greenfield, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] LaForce C, Journeay GE, Miller SD, Silvey MJ, Wu W, Lee LA, Chylack LT Jr. Ocular safety of fluticasone furoate nasal spray in patients with perennial allergic rhinitis: a 2-year study. Ann Allergy Asthma Immunol. 2013 Jul;111(1):45-50. doi: 10.1016/j.anai.2013.04.013. Epub 2013 May 12. PMID 23806459
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: FFR110537 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: FFR110537 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: FFR110537 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: FFR110537 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: FFR110537 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: FFR110537 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: FFR110537 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: The matching placebo nasal spray containing only fluticasone furoate (FF) vehicle was self-administered as two sprays per nostril each morning once daily (QD) for 104 weeks.
- FF 110 mcg QD: FF nasal spray aqueous suspension contained 0.05% micronized FF. Each spray contained approximately 27.5 micrograms (mcg) of FF; participants self-administered two sprays per nostril each morning QD for a total dose of 110 mcg for 104 weeks.
Period: Overall Study
Arm/Group | Placebo | FF 110 mcg QD
Started | 182 | 368
Completed | 104 | 199
Not Completed | 78 | 169
Not completed — Adverse Event | 12 | 23
Not completed — Lack of Efficacy | 2 | 0
Not completed — Protocol Violation | 38 | 76
Not completed — Met Protocol-defined Stopping Criteria | 3 | 4
Not completed — Lost to Follow-up | 1 | 6
Not completed — Physician Decision | 2 | 6
Not completed — Withdrawal by Subject | 19 | 53
Not completed — Did Not Receive Study Drug | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | FF 110 mcg QD | Total
Number analyzed (Participants) | 181 | 367 | 548
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline Characteristics were collected in members of the Intent-to-Treat (ITT) Population, comprised of all participants who were randomized and received at least one dose of double-blind study drug. One participant in the placebo group and one participant in the FF 110 mcg QD group did not receive any study drug and were thus not included in the ITT Population.
  Years | 38.0 (13.34) | 37.0 (13.48) | 37.4 (13.43)
Gender [Count of Participants; unit: Participants] — Baseline Characteristics were collected in members of the Intent-to-Treat (ITT) Population, comprised of all participants who were randomized and received at least one dose of double-blind study drug. One participant in the placebo group and one participant in the FF 110 mcg QD group did not receive any study drug and were thus not included in the ITT Population.
  Participants
    Female | 116 | 255 | 371
    Male | 65 | 112 | 177
Race/Ethnicity, Customized [Number; unit: participants] — Baseline Characteristics were collected in members of the Intent-to-Treat (ITT) Population, comprised of all participants who were randomized and received at least one dose of double-blind study drug. One participant in the placebo group and one participant in the FF 110 mcg QD group did not receive any study drug and were thus not included in the ITT Population.
  participants
    African American/African Heritage | 29 | 50 | 79
    American Indian or Alaska Native | 1 | 4 | 5
    Central/South Asian Heritage | 0 | 1 | 1
    Japanese/East Asian/South East Asian Heritage | 2 | 6 | 8
    Mixed Asian Heritage | 0 | 1 | 1
    Native Hawaiian or other Pacific Islander | 2 | 2 | 4
    White | 146 | 303 | 449
    African American/African Heritage & White | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Proportion (CU) of Participants (Par.) With an Event, as Measured as a Percentage, for Posterior Subcapsular Opacity (P)
Description: An event for P (opacity in the lens positioned just anterior to the posterior lens capsule and characterized by the posterior migration of lens epithelial cells from the lens bow) is defined as an increase of >=0.3 from baseline in Lens Opacities Classification System, Version III (LOCS III; system used for the grading and comparison of cataract severity and type based on standard color photographic transparencies) grade for P (range=0.1 [lens clear] to 5.9 [lens unclear]), in either eye. Data represent the Kaplan-Meier estimate for the CU of par. with an event of P based on a lifetest table.
Time Frame: Baseline; Weeks 12, 24, 36, 52, 64, 76, 88, and 104
Population: ITT Population. All participants (par.) with post-baseline ophthalmic examination data were included in the analysis for this endpoint. Par. without post-baseline ophthalmic exam data were censored at the randomization data. Par. who completed the study without an event for P or were discontinued for reasons other than an event for P were censored.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | FF 110 mcg QD
Number analyzed (Participants) | 168 | 344
Percentage of participants
  Week 12 | 0.60 | 0.88
  Week 24 | 1.24 | 1.84
  Week 36 | 1.93 | 2.56
  Week 52 | 2.68 | 3.72
  Week 64 | 2.68 | 3.72
  Week 76 | 2.68 | 3.72
  Week 88 | 2.68 | 4.59
  Week 104 | 2.68 | 5.09
Statistical Analysis 1: Comparison: Placebo vs FF 110 mcg QD; Test type: Superiority or Other; p = 0.395, Wald Chi-square — Wald Chi-Square test based on a proportional hazards model adjusting for age and baseline value

2. Primary Outcome: Cumulative Proportion of Participants, as Measured as a Percentage, With an Intraocular Pressure (IOP) Event
Description: An event for IOP is defined as an increase of 7 millimeters of mercury (mm Hg) or greater from baseline in IOP, in either eye, using Goldmann Applanation Tonometry (GAT). GAT is a commonly used method of determining approximate intraocular pressure. The data below represent the Kaplan-Meier estimate for the cumulative proportion of participants with an IOP event based on a lifetest table.
Time Frame: Baseline; Weeks 12, 24, 36, 52, 64, 76, 88, and 104
Population: ITT Population. All participants with post-baseline ophthalmic examination data were included in the analysis for this endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | FF 110 mcg QD
Number analyzed (Participants) | 168 | 344
percentage of participants
  Week 12 | 0.00 | 0.00
  Week 24 | 0.00 | 0.32
  Week 36 | 0.00 | 0.32
  Week 52 | 0.00 | 0.71
  Week 64 | 0.00 | 1.12
  Week 76 | 0.00 | 1.98
  Week 88 | 0.84 | 1.98
  Week 104 | 0.84 | 2.96
Statistical Analysis 1: Comparison: Placebo vs FF 110 mcg QD; Test type: Superiority or Other; p = 0.342, Wald Chi-square — Wald Chi-Square test based on a proportional hazards model adjusting for age and baseline value

3. Secondary Outcome: Change From Baseline in LOCS III Posterior Subcapsular Opacity at Week 52 and Week 104
Description: An event for P (opacity in the lens positioned just anterior to the posterior lens capsule and characterized by the posterior migration of lens epithelial cells from the lens bow) is defined as an increase of >=0.3 from baseline in LOCS III (system used for the grading and comparison of cataract severity and type based on standard color photographic transparencies) grade for P (range=0.1 [lens clear] to 5.9 [lens unclear]), in either eye. Change from baseline was calculated by subtracting the baseline value from the Week 52 and Week 104 value.
Time Frame: Baseline, Week 52, and Week 104
Population: ITT Population. The number analyzed reflects those participants remaining in the study and contributing data at the indicated time points.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | FF 110 mcg QD
Number analyzed (Participants) | 130 | 198
scores on a scale
  Left eye, Week 52; n=130, 251 | 0.00 (0.042) | 0.00 (0.063)
  Left eye, Week 104; n=104, 198 | 0.00 (0.039) | 0.00 (0.083)
  Right eye, Week 52; n=130, 251 | 0.00 (0.057) | 0.00 (0.061)
  Right eye, Week 104; n=104, 198 | 0.00 (0.042) | -0.01 (0.068)

4. Secondary Outcome: Number of Participants With the Indicated Change From Baseline in LOCS III Posterior Subcapsular Opacity by Increments of 0.1 at Weeks 52 and 104
Description: An event for P is defined as an increase of >=0.3 from baseline in LOCS III (classification system based on standard color photographic transparencies) grade for P (range=0.1 [lens clear] to 5.9 [lens unclear]), in either eye. Change from baseline was calculated by subtracting the baseline value from the Week 52 and Week 104 value.
Time Frame: Baseline, Week 52, and Week 104
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Placebo | FF 110 mcg QD
Number analyzed (Participants) | 130 | 251
participants
  Left eye, Week 52, <-0.3; n=130, 251 | 0 | 0
  Left eye, Week 52, -0.3; n=130, 251 | 0 | 0
  Left eye, Week 52, -0.2; n=130, 251 | 2 | 5
  Left eye, Week 52, -0.1; n=130, 251 | 3 | 13
  Left eye, Week 52, 0; n=130, 251 | 121 | 218
  Left eye, Week 52, 0.1; n=130, 251 | 3 | 12
  Left eye, Week 52, 0.2; n=130, 251 | 0 | 0
  Left eye, Week 52, 0.3; n=130, 251 | 1 | 2
  Left eye, Week 52, 0.4; n=130, 251 | 0 | 0
  Left eye, Week 52, 0.5; n=130, 251 | 0 | 0
  Left eye, Week 52, 0.6; n=130, 251 | 0 | 1
  Left eye, Week 52, 0.7; n=130, 251 | 0 | 0
  Left eye, Week 52, 0.8; n=130, 251 | 0 | 0
  Left eye, Week 52, >=0.9; n=130, 251 | 0 | 0
  Left eye, Week 52, >=0.3; n=130, 251 | 1 | 3
  Left eye, Week 52, >=0.5; n=130, 251 | 0 | 1
  Left eye, Week 52, >=1.0; n=130, 251 | 0 | 0
  Right eye, Week 52, <-0.3; n=130, 251 | 0 | 0
  Right eye, Week 52, -0.3; n=130, 251 | 1 | 0
  Right eye, Week 52, -0.2; n=130, 251 | 1 | 5
  Right eye, Week 52, -0.1; n=130, 251 | 0 | 10
  Right eye, Week 52, 0; n=130, 251 | 122 | 218
  Right eye, Week 52, 0.1; n=130, 251 | 4 | 13
  Right eye, Week 52, 0.2; n=130, 251 | 0 | 2
  Right eye, Week 52, 0.3; n=130, 251 | 1 | 1
  Right eye, Week 52, 0.4; n=130, 251 | 1 | 2
  Right eye, Week 52, 0.5; n=130, 251 | 0 | 0
  Right eye, Week 52, 0.6; n=130, 251 | 0 | 0
  Right eye, Week 52, 0.7; n=130, 251 | 0 | 0
  Right eye, Week 52, 0.8; n=130, 251 | 0 | 0
  Right eye, Week 52, >=0.9; n=130, 251 | 0 | 0
  Right eye, Week 52, >=0.3; n=130, 251 | 2 | 3
  Right eye, Week 52, >=0.5; n=130, 251 | 0 | 0
  Right eye, Week 52, >=1.0; n=130, 251 | 0 | 0
  Left eye, Week 104, <-0.3; n=104, 198 | 0 | 0
  Left eye, Week 104, -0.3; n=104, 198 | 0 | 0
  Left eye, Week 104, -0.2; n=104, 198 | 2 | 5
  Left eye, Week 104, -0.1; n=104, 198 | 3 | 11
  Left eye, Week 104, 0; n=104, 198 | 94 | 175
  Left eye, Week 104, 0.1; n=104, 198 | 5 | 5
  Left eye, Week 104, 0.2; n=104, 198 | 0 | 0
  Left eye, Week 104, 0.3; n=104, 198 | 0 | 0
  Left eye, Week 104, 0.4; n=104, 198 | 0 | 0
  Left eye, Week 104, 0.5; n=104, 198 | 0 | 0
  Left eye, Week 104, 0.6; n=104, 198 | 0 | 1
  Left eye, Week 104, 0.7; n=104, 198 | 0 | 0
  Left eye, Week 104, 0.8; n=104, 198 | 0 | 1
  Left eye, Week 104, >=0.9; n=104, 198 | 0 | 0
  Left eye, Week 104, >=0.3; n=104, 198 | 0 | 2
  Left eye, Week 104, >=0.5; n=104, 198 | 0 | 2
  Left eye, Week 104, >=1.0; n=104, 198 | 0 | 0
  Right eye, Week 104, <-0.3; n=104, 198 | 0 | 0
  Right eye, Week 104, -0.3; n=104, 198 | 1 | 0
  Right eye, Week 104, -0.2; n=104, 198 | 1 | 5
  Right eye, Week 104, -0.1; n=104, 198 | 2 | 14
  Right eye, Week 104, 0; n=104, 198 | 97 | 174
  Right eye, Week 104, 0.1; n=104, 198 | 3 | 2
  Right eye, Week 104, 0.2; n=104, 198 | 0 | 2
  Right eye, Week 104, 0.3; n=104, 198 | 0 | 0
  Right eye, Week 104, 0.4; n=104, 198 | 0 | 0
  Right eye, Week 104, 0.5; n=104, 198 | 0 | 0
  Right eye, Week 104, 0.6; n=104, 198 | 0 | 0
  Right eye, Week 104, 0.7; n=104, 198 | 0 | 1
  Right eye, Week 104, 0.8; n=104, 198 | 0 | 0
  Right eye, Week 104, >=0.9; n=104, 198 | 0 | 0
  Right eye, Week 104, >=0.3; n=104, 198 | 0 | 1
  Right eye, Week 104, >=0.5; n=104, 198 | 0 | 1
  Right eye, Week 104, >=1.0; n=104, 198 | 0 | 0

5. Secondary Outcome: Change From Baseline in LOCS III Cortical Opacity (C) at Week 52 and Week 104
Description: An event for C (an opacity starting at the outer edge of the lens and progressing toward the center) is defined as an increase of >=0.3 from baseline in LOCS III (system used for the grading and comparison of cataract severity and type based on standard color photographic transparencies) grade for C (range=0.1 [lens clear] to 5.9 [lens unclear]), in either eye. Change from baseline was calculated by subtracting the baseline value from the Week 52 and Week 104 value.
Time Frame: Baseline, Week 52, and Week 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | FF 110 mcg QD
Number analyzed (Participants) | 130 | 251
scores on a scale
  Left eye, Week 52; n=130, 251 | 0.01 (0.210) | 0.00 (0.113)
  Left eye, Week 104; n=104, 198 | 0.02 (0.210) | 0.01 (0.186)
  Right eye, Week 52; n=130, 251 | -0.01 (0.229) | 0.00 (0.154)
  Right eye, Week 104; n=104, 198 | 0.02 (0.187) | 0.01 (0.186)

6. Secondary Outcome: Number of Participants With the Indicated Change From Baseline in Cortical Opacity by Increment Categories of >=0.3, >=0.5, and >=1.0 at Weeks 52 and 104
Description: as for outcome 5
Time Frame: Baseline, Week 52, and Week 104
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Placebo | FF 110 mcg QD
Number analyzed (Participants) | 130 | 251
participants
  Left eye, Week 52, >=0.3; n=130, 251 | 4 | 4
  Left eye, Week 52, >=0.5; n=130, 251 | 1 | 0
  Left eye, Week 52, >=1.0; n=130, 251 | 1 | 0
  Right eye, Week 52, >=0.3; n=130, 251 | 3 | 8
  Right eye, Week 52, >=0.5; n=130, 251 | 1 | 2
  Right eye, Week 52, >=1.0; n=130, 251 | 1 | 0
  Left eye, Week 104, >=0.3; n=104, 198 | 6 | 10
  Left eye, Week 104, >=0.5; n=104, 198 | 3 | 4
  Left eye, Week 104, >=1.0; n=104, 198 | 1 | 1
  Right eye, Week 104, >=0.3; n=104, 198 | 3 | 10
  Right eye, Week 104, >=0.5; n=104, 198 | 2 | 4
  Right eye, Week 104, >=1.0; n=104, 198 | 1 | 2

7. Secondary Outcome: Change From Baseline in LOCS III Nuclear Opacity (NO) at Week 52 and Week 104
Description: Nuclear opacity refers to the opacity in the central nucleus of the eye.The range for NO is 0.1 (no opacity) to 6.9 (maximum opacity). Change from baseline in NO was calculated by subtracting the baseline value from the Week 52 or Week 104 value.
Time Frame: Baseline, Week 52, and Week 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | FF 110 mcg QD
Number analyzed (Participants) | 130 | 251
scores on a scale
  Left eye, Week 52; n=130, 251 | 0.12 (0.498) | 0.06 (0.495)
  Left eye, Week 104; n=104, 198 | 0.21 (0.538) | 0.10 (0.506)
  Right eye, Week 52; n=130, 251 | 0.12 (0.511) | 0.06 (0.492)
  Right eye, Week 104; n=104, 198 | 0.21 (0.550) | 0.09 (0.531)

8. Secondary Outcome: Change From Baseline in Nuclear Color (NC) at Week 52 and Week 104
Description: Nuclear color is associated with the force required to compress a lens to 75% of its original depth. The range for NC is 0.1 (no opacity) to 6.9 (maximum opacity). Change from baseline in NC was calculated by subtracting the baseline value from the Week 52 or Week 104 value.
Time Frame: Baseline, Week 52, and Week 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | FF 110 mcg QD
Number analyzed (Participants) | 130 | 251
scores on a scale
  Left eye, Week 52; n=130, 251 | 0.14 (0.432) | 0.09 (0.402)
  Left eye, Week 104; n=104, 198 | 0.21 (0.454) | 0.13 (0.465)
  Right eye, Week 52; n=130, 251 | 0.16 (0.422) | 0.09 (0.410)
  Right eye, Week 104; n=104, 198 | 0.22 (0.452) | 0.13 (0.469)

9. Secondary Outcome: Change From Baseline in Intraocular Pressure (IOP) at Weeks 52 and 104
Description: An event for IOP is defined as an increase of 7 mm Hg or greater from baseline in IOP, in either eye, using Goldmann Applanation Tonometry. Participants without post-baseline ophthalmic exam data were censored at the randomization date. Change from baseline was calculated by subtracting the baseline value from the Week 52 or Week 104 value.
Time Frame: Baseline, Week 52, and Week 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Placebo: An event for IOP is defined as an increase of 7 mm Hg or greater from baseline in IOP, in either eye, using Goldmann Applanation Tonometry. Participants without post-baseline ophthalmic exam data were censored at the randomization date. Change from baseline was calculated by subtracting the baseline value from the Week 52 or Week 104 value.
Arm/Group | Placebo | FF 110 mcg QD
Number analyzed (Participants) | 130 | 251
mm Hg
  Left eye, Week 52; n=130, 251 | -0.5 (2.04) | -0.3 (2.26)
  Left eye, Week 104; n=104, 198 | -0.8 (1.98) | -0.6 (2.41)
  Right eye, Week 52; n=130, 251 | -0.7 (2.08) | -0.4 (2.33)
  Right eye, Week 104; n=104, 198 | -1.0 (2.17) | -0.7 (2.55)

10. Secondary Outcome: Number of Participants With the Indicated Change From Baseline in Intraocular Pressure (IOP) by Increments of 1 mm Hg at Week 52
Description: An event for IOP is defined as an increase of 7 mm Hg or greater from baseline in IOP, in either eye, using Goldmann Applanation Tonometry. Participants without post-baseline ophthalmic exam data were censored at the randomization date. Change from baseline was calculated by subtracting the baseline value from the Week 52 value.
Time Frame: Baseline and Week 52
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Placebo | FF 110 mcg QD
Number analyzed (Participants) | 130 | 251
participants
  Left eye, IOP = <-10 to -9 | 1 | 0
  Left eye, IOP = -8 | 0 | 0
  Left eye, IOP = -7 | 0 | 2
  Left eye, IOP = -6 | 0 | 0
  Left eye, IOP = -5 | 3 | 3
  Left eye, IOP = -4 | 5 | 12
  Left eye, IOP = -3 | 9 | 19
  Left eye, IOP = -2 | 18 | 40
  Left eye, IOP = -1 | 22 | 40
  Left eye, IOP = 0 | 36 | 50
  Left eye, IOP = 1 | 20 | 30
  Left eye, IOP = 2 | 7 | 24
  Left eye, IOP = 3 | 5 | 19
  Left eye, IOP = 4 | 4 | 7
  Left eye, IOP = 5 | 0 | 3
  Left eye, IOP = 6 | 0 | 2
  Left eye, IOP = 7 | 0 | 0
  Left eye, IOP = 8 | 0 | 0
  Left eye, IOP = 9 | 0 | 0
  Left eye, IOP >= 7 | 0 | 0
  Left eye, IOP >= 10 | 0 | 0
  Left eye, IOP >= 15 | 0 | 0
  Right eye, IOP = <-10 to -9 | 0 | 0
  Right eye, IOP = -8 | 0 | 1
  Right eye, IOP = -7 | 2 | 0
  Right eye, IOP = -6 | 0 | 1
  Right eye, IOP = -5 | 2 | 4
  Right eye, IOP = -4 | 7 | 14
  Right eye, IOP = -3 | 9 | 23
  Right eye, IOP = -2 | 25 | 43
  Right eye, IOP = -1 | 22 | 34
  Right eye, IOP = 0 | 28 | 46
  Right eye, IOP = 1 | 16 | 31
  Right eye, IOP = 2 | 13 | 27
  Right eye, IOP = 3 | 3 | 14
  Right eye, IOP = 4 | 2 | 8
  Right eye, IOP = 5 | 1 | 2
  Right eye, IOP = 6 | 0 | 3
  Right eye, IOP = 7 | 0 | 0
  Right eye, IOP = 8 | 0 | 0
  Right eye, IOP = 9 | 0 | 0
  Right eye, IOP >= 7 | 0 | 0
  Right eye, IOP >= 10 | 0 | 0
  Right eye, IOP >= 15 | 0 | 0

11. Secondary Outcome: Number of Participants With the Indicated Change From Baseline in Intraocular Pressure (IOP) by Increments of 1 mm Hg at Week 104
Description: An event for IOP is defined as an increase of 7 mm Hg or greater from baseline in IOP, in either eye, using Goldmann Applanation Tonometry. Participants without post-baseline ophthalmic exam data were censored at the randomization date. Change from baseline in IOP was calculated by subtracting the baseline value from the Week 104 value.
Time Frame: Baseline and Week 104
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Placebo | FF 110 mcg QD
Number analyzed (Participants) | 104 | 198
participants
  Left eye, IOP = <-10 to -9 | 0 | 0
  Left eye, IOP = -8 | 0 | 1
  Left eye, IOP = -7 | 0 | 0
  Left eye, IOP = -6 | 2 | 3
  Left eye, IOP = -5 | 0 | 7
  Left eye, IOP = -4 | 6 | 10
  Left eye, IOP = -3 | 15 | 19
  Left eye, IOP = -2 | 17 | 31
  Left eye, IOP = -1 | 15 | 32
  Left eye, IOP = 0 | 21 | 32
  Left eye, IOP = 1 | 19 | 30
  Left eye, IOP = 2 | 5 | 16
  Left eye, IOP = 3 | 3 | 7
  Left eye, IOP = 4 | 0 | 6
  Left eye, IOP = 5 | 1 | 2
  Left eye, IOP = 6 | 0 | 1
  Left eye, IOP = 7 | 0 | 1
  Left eye, IOP = 8 | 0 | 0
  Left eye, IOP = 9 | 0 | 0
  Left eye, IOP >= 7 | 0 | 1
  Left eye, IOP >= 10 | 0 | 0
  Left eye, IOP >= 15 | 0 | 0
  Right eye, IOP = <-10 to -9 | 0 | 0
  Right eye, IOP = -8 | 0 | 1
  Right eye, IOP = -7 | 0 | 2
  Right eye, IOP = -6 | 2 | 1
  Right eye, IOP = -5 | 5 | 7
  Right eye, IOP = -4 | 4 | 15
  Right eye, IOP = -3 | 10 | 17
  Right eye, IOP = -2 | 24 | 32
  Right eye, IOP = -1 | 21 | 22
  Right eye, IOP = 0 | 12 | 46
  Right eye, IOP = 1 | 16 | 23
  Right eye, IOP = 2 | 6 | 13
  Right eye, IOP = 3 | 1 | 8
  Right eye, IOP = 4 | 1 | 5
  Right eye, IOP = 5 | 1 | 2
  Right eye, IOP = 6 | 1 | 2
  Right eye, IOP = 7 | 0 | 2
  Right eye, IOP = 8 | 0 | 0
  Right eye, IOP = 9 | 0 | 0
  Right eye, IOP >= 7 | 0 | 2
  Right eye, IOP >= 10 | 0 | 0
  Right eye, IOP >= 15 | 0 | 0

12. Secondary Outcome: Change From Baseline in Logarithm of the Minimum Angle of Resolution (LogMAR) Visual Acuity (VA) Using Early Treatment Diabetic Retinopathy Study (ETDRS) Charts at Week 52 and Week 104
Description: ETDRS charts are used to measure VA (the ability to resolve fine image details). Participants must have had a best-corrected distance VA of =< 0.18 on the LogMAR scale using ETDRS charts in both eyes measured separately. The LogMAR scale (expressed as the [decadic] logarithm of the minimum angle of resolution [range from +1.00 to -0.30]) converts the geometric sequence of a traditional chart to a linear scale. It measures VA loss; positive values indicate vision loss, whereas negative values denote normal or better VA. A lower LogMAR value indicates better VA.
Time Frame: Baseline, Week 52, and Week 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | FF 110 mcg QD
Number analyzed (Participants) | 130 | 251
scores on a scale
  Left eye, Week 52; n=130, 251 | -0.027 (0.0729) | -0.013 (0.0778)
  Left eye, Week 104; n=104, 198 | -0.035 (0.0740) | -0.023 (0.0858)
  Right eye, Week 52; n=130, 251 | -0.023 (0.0810) | -0.014 (0.0852)
  Right eye, Week 104; n=104, 198 | -0.025 (0.0992) | -0.024 (0.0899)

13. Secondary Outcome: Percent Change From Baseline in the Funduscopic Horizontal Cup-to-disc Ratio at Week 104
Description: The funduscopic horizontal cup-to-risk ratio assesses the progression of glaucoma. Percent change from baseline in funduscopic horizontal cup-to-disc ratio at Week 104 was calculated by substracting the baseline value from the Week 104 value (both expressed as a percent). The cup-to-disc ratio compares the diameter of the "cup" portion of the optic disc with the total diameter of the optic disc. A large cup-to-disc ratio may imply glaucoma or other pathology.
Time Frame: Baseline and Week 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | FF 110 mcg QD
Number analyzed (Participants) | 104 | 198
percent change
  Left eye | 0.0 (7.23) | 0.7 (7.58)
  Right eye | 0.0 (7.31) | 0.0 (7.39)

14. Secondary Outcome: Change From Baseline in the Daily Reflective Total Nasal Symptom Score (rTNSS) for the Indicated Study Periods
Description: rTNSS was evaluated on a 4-point categorical scale (sum of the scores for rhinorrhea, nasal congestion, nasal itching, and sneezing; range=0-12). The data collected were used as a measure for treatment compliance. The scores on the scale were based on the severity of each nasal symptom: 0=none (symptom is not present); 1=mild (sign/symptom is clearly present but minimal awareness; easily tolerated); 2=moderate (definite awareness of sign/symptom that is bothersome but tolerable); 3=severe (sign/symptom is hard to tolerate; causes interference with activities of daily living and/or sleeping).
Time Frame: Baseline, Weeks 1 to 26, Weeks 27 to 52, Weeks 53 to 78, and Weeks 79 to 104
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | FF 110 mcg QD
Number analyzed (Participants) | 181 | 367
scores on a scale
  Week 1 to 26 | -2.12 (0.17) | -3.19 (0.12)
  Week 27 to 52 | -2.52 (0.21) | -3.86 (0.15)
  Week 53 to 78 | -2.56 (0.23) | -3.89 (0.16)
  Week 79 to 104 | -2.59 (0.25) | -4.10 (0.18)
  Week 1 to 104 | -2.30 (0.18) | -3.45 (0.13)

ADVERSE EVENTS:
Arm/Group | Placebo | FF 110 mcg QD
Serious Adverse Events (participants affected / at risk) | 7/181 | 12/367
Other Adverse Events (participants affected / at risk) | 97/181 | 232/367
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=181) | FF 110 mcg QD (N=367)
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 2
Intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Blood pressure increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=181) | FF 110 mcg QD (N=367)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 34 | 123
Sinusitis (Infections and infestations) | 31 | 47
Upper respiratory tract infection (Infections and infestations) | 29 | 52
Nasopharyngitis (Infections and infestations) | 17 | 44
Influenza (Infections and infestations) | 16 | 25
Viral upper respiratory tract infection (Infections and infestations) | 12 | 27
Headache (Nervous system disorders) | 13 | 29
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 23
Bronchitis (Infections and infestations) | 8 | 31
Acute sinusitis (Infections and infestations) | 7 | 20
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 3 | 30
Nasal septum ulceration (Respiratory, thoracic and mediastinal disorders) | 6 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.